CLINICAL TRIAL: NCT02396589
Title: Feasibility of a Novel Intervention to Improve Participation After Stroke
Brief Title: Community Participation Transition After Stroke
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Susan Stark, Assisstant Professor of Neurology and Occupational Therapy, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCMRR 1611R03HD079841-01A1
Record Dates: First submitted 2015-03-05; First posted 2015-03-24 (Estimated); Results first posted 2024-04-12 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: stroke rehabilitation; barriers to independence; environmental support
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education Group (Active Comparator): Participants in the Education group receive five 90 minute tailored stroke education sessions in the home.
  Interventions: Behavioral: Education Group
- Home Modifications Group (Experimental): Participants in the treatment group receive a home assessment and home modifications tailored to functional abilities (pre discharge) and then five 90 minute occupational therapy treatment sessions at home (post discharge) to improve functional abilities and community participation.
  Interventions: Behavioral: Home Modifications Group

INTERVENTIONS:
Behavioral: Education Group — Attention will be provided to the control group to ensure they experience the same effects of time and attention but no effect on the outcome of interest.
  Arms: Education Group
Behavioral: Home Modifications Group — The standardized components include assessment, identification of five problematic activities (and environmental barriers), identification of three solutions (for each problem), implementation of a solution set selected by the participant, training, and active practice of daily activities in one's own home and community.
  Arms: Home Modifications Group

SUMMARY:
Stroke is one of the most serious, disabling health conditions in the United States. Patients who undergo rehabilitation treatment for stroke have a high rate of disability. Poor outcomes for many persons with stroke may be low because of incomplete treatment. The investigators will conduct a randomized controlled trial and a process evaluation to examine the feasibility, safety, and preliminary efficacy of an enhanced rehabilitation transition program, Community Participation Transition after Stroke (COMPASS), designed to bridge inpatient rehabilitation and the home to support the performance of everyday activities.

DETAILED DESCRIPTION:
We propose an enhanced rehabilitation transition program: Community Participation Transition after Stroke (COMPASS) is a compensatory intervention consisting of one pre-discharge and five post-discharge home visits by an occupational therapist to supplement usual care. This intervention is focused on resolving barriers to independence in daily activities and participation using environmental support and active practice of daily activities in an individual's real home (versus an idealized clinical setting). This is a new combination of evidence-based compensatory treatments delivered in a novel treatment setting (transition to home). Our long-term goal is the development of an effective intervention for a transition home designed to prevent excess disability for people living with stroke that could have an immediate effect and high public health significance.16

We will recruit 40 patients currently undergoing inpatient rehabilitation (IR) for ischemic stroke from longitudinal studies of stroke at Washington University School of Medicine (WUSM) and randomize them to receive six additional sessions of the enhanced rehabilitation transition program or attention control. Exploratory participation outcomes will be assessed by blinded evaluators at baseline, 6 months, 9 months, and 12 months after stroke.

We will test the central hypothesis that COMPASS will be acceptable, feasible, and superior to attention control on measures of participation and daily activity performance at 6 months after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. ≥45 years old
2. acute ischemic stroke, verified by a neurologist
3. baseline National Institutes of Health Stroke Scale (NIHSS) ≥8
4. independent in activities of daily living prior to stroke (premorbid Rankin score of ≤2)
5. plan to discharge to home

Exclusion Criteria:

1. severe terminal systemic disease that limits life expectancy to <6 months
2. previous disorder (e.g., dementia) that makes interpretation of the self-rated scales difficult or a Short Blessed Test (SBT) score of ≥9 (indicating significant cognitive impairment)
3. moderate to severe aphasia, as determined by the NIHSS Best Language rating of ≥2
4. residence in a congregate living facility
5. not eligible for a therapeutic pass

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Stark, PhD, Principal Investigator — Washington University School of Medicine, Program in Occupational Therapy
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Intervention
Arm/Group | Education Group | Home Modifications Group
Started | 6 | 9
Completed | 5 | 9
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: 6 Month Follow-up
Arm/Group | Education Group | Home Modifications Group
Started | 5 | 9
Completed | 5 | 8
Not Completed | 0 | 1
Not completed — change in health status | 0 | 1
Period: 9 Month Follow-up
Arm/Group | Education Group | Home Modifications Group
Started | 5 | 8
Completed | 5 | 7
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: 12 Month Follow up
Arm/Group | Education Group | Home Modifications Group
Started | 5 | 7
Completed | 5 | 5
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Group | Home Modifications Group | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (8.21) | 66.9 (7.96) | 66.0 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15
Length of Stay in Inpatient Rehabilitation [Mean (Standard Deviation); unit: days] — Length of stay is a clinical metric that measures the length of time elapsed between a patient's date of admission and discharge.
  days | 16.7 (53.5) | 24.1 (7.9) | 21.1 (7.8)
Stroke Impact Scale (SIS) Total [Mean (Standard Deviation); unit: units on a scale] — The Stroke Impact Scale (SIS) is a stroke-specific, self-report, health status measure. We are using the 10 items from the Activities of Daily Living / Instrumental Activities of Daily Living (ADL/IADL) domain. Clients also rate their overall recovery on a scale of 0 - 100, 0 indicating no recovery, 100 full recovery.
  units on a scale | 40.83 (22.00) | 38.33 (21.79) | 39.33 (21.12)
Reintegration to Normal Living Index (RNLI) [Mean (Standard Deviation); unit: units on a scale] — The RNLI measure the extent to which a person is able to resume normal life activities after illness or injury. The 11 items questionnaire asks about one's daily functioning and perception of self. Questions are scored on a scale of 1 to 10, with a 1 indicating the statement "does not describe my situation" and a 10 indicating the statement "fully describes my situation". Scores are summed for a total score out of 110 points which is then converted to an adjusted score with a range of 0-100. A higher score indicates higher attainment of normal levels of living. Scores reported are adjusted.
  units on a scale | 62.88 (22.24) | 52.73 (18.87) | 56.79 (20.12)
SIS Activity of Daily Living (ADL) Subscale [Mean (Standard Deviation); unit: units on a scale] — The Stroke Impact Scale (SIS) is a stroke-specific, self-report, health status measure. We are using the 10 items from the Activities of Daily Living / Instrumental Activities of Daily Living (ADL/IADL) domain. Each item is rated using a 5-point Likert scale, with a 1 indicating an inability to complete the activity and a 5 indicating no difficulty experienced at all. Domain scores range from 0-100 and are calculated using the following equation = [(Mean item score - 1) / 5-1 ] x 100.
  units on a scale | 52.83 (15.03) | 37.11 (17.09) | 43.4 (17.64)
In-Home Occupational Performance Measure (I-HOPE) Performance [Mean (Standard Deviation); unit: units on a scale] — The I-HOPE is a multi-step assessment that evaluates performance of older adults doing 42 activities in the home. It measures current activity patterns of participants, identifies activities that are difficult but important to them, and identifies environmental barriers that influence those activities. Participants rate their performance of top 10 desired activities on a scale of 1-5, with 1=no performance and 5=perfect performance. A sum (score range 10-50) and mean score (range 1-5) are calculated for all 10 activities. Scores reported are sum scores. Higher sum scores= better performance.
  units on a scale | 16.00 (7.72) | 21.22 (5.76) | 19.13 (6.88)
I-HOPE Satisfaction [Mean (Standard Deviation); unit: units on a scale] — The I-HOPE is a multi-step assessment evaluating performance of older adults for 42 activities in the home. It measures activity patterns of participants, identifies activities that are difficult but important to them, and identifies environmental barriers influencing those activities. Participants rate their satisfaction with their ability to perform each problematic activity on a scale of 1-5, with 1=not satisfied at all, and 5= totally satisfied. A sum (range 10-50) and mean score (range 1-5) are calculated for all 10 activities. Sum scores are reported. Higher scores=greater satisfaction.
  units on a scale | 16.67 (9.40) | 19.33 (5.94) | 18.27 (7.31)
I-HOPE Environmental Barriers [Mean (Standard Deviation); unit: barrier score] — The I-HOPE is a multi-step assessment that evaluates the performance of older adults doing 42 activities in the home. The I-HOPE measures current activity patterns of participants, identifies activities that are difficult but important, and identifies environmental barriers that influence activity performance. The barrier scores is an objective score of the impact of the environment on ability to perform daily activities. Barriers scores range from 0, no impact on performance to 5, total impact on performance. Higher barrier scores indicate worse performance. Barriers scores are summed.
  barrier score | 58.67 (35.01) | 85.44 (22.47) | 74.73 (30.18)

OUTCOME MEASURES:

1. Primary Outcome: Rate and Severity of Falls (Calculated With an Algorithm)
Description: We will explore the safety of the intervention by determining the rate and severity of falls (calculated with an algorithm). Scores are as follows: 0, those with no falls, 1, those with one fall without serious injury, 2, those with at least two falls without serious injury, and 3, those with one or more falls causing serious injury. Maximum score of three indicates an increased severity of fall. We will compare the difference in scores between groups using t-tests.
Time Frame: 12 months
Population: 15 participants were randomized (treatment group n=9 and education group n=6). 12 participants were included in this analysis. One participant in the education group was not able to finish education visits and was excluded from the analysis. Two participants in the treatment group were lost to follow up (drop out due to change in health n=1, drop out due to death n=1), and were excluded from analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Group | Home Modifications Group
Number analyzed (Participants) | 5 | 7
score on a scale | 2 (.316) | 2 (.00)

2. Secondary Outcome: Intervention Dose (Minutes)
Description: The does of the intervention as measured in minutes received by both groups. The number of minutes reported is the average of the total for each participant in each group.
Time Frame: 2 months
Population: A total of 14 participants were analyzed. One participant in the education group was not able to finish the education visits and was excluded from this analysis.
Measure: Mean (Standard Deviation); unit: number of treatment minutes
Arm/Group | Education Group | Home Modifications Group
Number analyzed (Participants) | 5 | 9
number of treatment minutes | 354.8 (120.1) | 365 (108.3)

3. Secondary Outcome: Health Care Utilization, Number of Emergency Department Visits
Description: We analyzed health care utilization by examining the number of emergency department visits, outpatient physical and occupational therapy visits, and doctor visits. The total number of each was calculated for each participant and the average is reported here.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Education Group | Home Modifications Group
Number analyzed (Participants) | 5 | 7
Number of visits
  Emergency Room Visits | .50 (.55) | .56 (.88)
  Outpatient physical therapy visits | 28.67 (34.72) | 26.11 (30.10)
  Outpatient occupational therapy visits | 36.00 (36.30) | 19.44 (24.14)
  Outpatient doctor visits | 10.33 (10.86) | 26.11 (30.10)

4. Secondary Outcome: Intervention Dose, Number of Treatment Sessions
Description: The does of the intervention as measured by amount of treatment minutes received by both groups. The total number of treatment sessions was calculated for each participant and the average is reported here.
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of treatment sessions
Arm/Group | Education Group | Home Modifications Group
Number analyzed (Participants) | 5 | 9
number of treatment sessions | 4.4 (1.3) | 5 (1)

5. Secondary Outcome: Health Care Utilization, Days of Hospitalization
Description: We analyzed health care utilization by examining the number of days participants in each group spent in the hospital. The total number of days was calculated for participants in each group and the average is reported here.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Education Group | Home Modifications Group
Number analyzed (Participants) | 5 | 7
days | 0 (0) | .67 (1.12)

6. Other Pre Specified Outcome: Intervention Adherence
Description: Adherence to the intervention will be measured by examine the number of recommendations implemented per recommendations suggested. Long-term adherence will be calculated as the number of recommendations used at 9 months per recommendations suggested.
Time Frame: 9 months
Population: 9 participants were randomized to the treatment group. 7 participants were included in this analysis. Two participants in the treatment group were lost to follow up (drop out due to change in health n=1, drop out due to death n=1), and were excluded from analysis.
Measure: Mean (Standard Deviation); unit: percentage of recommendations used
Arm/Group | Home Modifications Group
Number analyzed (Participants) | 7
percentage of recommendations used | 71.25 (31)

ADVERSE EVENTS:
Arm/Group | Education Group | Home Modifications Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 0/6 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Education Group (N=6) | Home Modifications Group (N=9)
Hospitalization (General disorders) | 0 (0) | 0 (0) — Participants were asked "How many hospitalizations have you had in the past 6 months?" and were able to self-report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No